CLINICAL TRIAL: NCT03996161
Title: Effect of Semi-sitting Position on Mask Ventilation in Anesthetized and Paralyzed Patients
Brief Title: Effect of Semi-sitting Position on Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019-1231
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Ventilation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine position (Active Comparator): After the induction of anesthesia, mask ventilation is performed in the supine position.
  Interventions: Other: patient position
- Semi-sitting position (Experimental): After the induction of anesthesia, mask ventilation is performed in the semi-sitting position.
  Interventions: Other: patient position

INTERVENTIONS:
Other: patient position — After the induction of anesthesia, mask ventilation is performed in the supine and semi-sitting position in a cross-over, randomized order.

SUMMARY:
We compare the effect on semi-sitting position on mask ventilation in anesthetized and paralyzed obese patients

ELIGIBILITY:
Inclusion Criteria:

* Obese patients undergoing general anesthesia

Exclusion Criteria:

* diseases or structural abnormalities in the upper airway
* those who were at risk of aspiration
* cardiovascular or respiratory diseases
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Expiratory tidal volume | 1 minute after the induction of anesthesia
  Expiratory tidal volume is assessed during mask ventilation in the supine and semi-sitting positions.

SECONDARY OUTCOMES:
Minute ventilation during mask ventilation in the supine and semi-sitting positions | 1 minute after anesthesia induction
  Minute ventilation is assessed during mask ventilation
The incidence of inadequate mask ventilation or dead space ventilation. | during mask ventilation
  The incidence of inadequate mask ventilation or dead space ventilation is recorded.
Peak inspiratory pressure | during mask ventilation
  Peak inspiratory pressure is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chang JE, Seol T, Hwang JY. Body position and the effectiveness of mask ventilation in anaesthetised paralysed obese patients: A randomised cross-over study. Eur J Anaesthesiol. 2021 Aug 1;38(8):825-830. doi: 10.1097/EJA.0000000000001473. PMID 33600105